CLINICAL TRIAL: NCT02720016
Title: An Integrative Technology Approach to Home-based Conjoint Therapy for PTSD
Brief Title: Cognitive-Behavioral Conjoint Therapy (CBCT) Project
Acronym: CBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2093-R; H150181 (Other: VA HRPP)
Record Dates: First submitted 2016-03-07; First posted 2016-03-25 (Estimated); Results first posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2021-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder; Marital Therapy; Veterans; Telemedicine; Couples
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study assessors are kept blind to the couple's randomly assigned treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CBCT-Home Based (CBCT-HB) (Experimental): Couples in CBCT-HB will receive 8 sessions of standardized Cognitive-Behavioral Conjoint Therapy (CBCT), a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning. The psychotherapy is administered over 8 to 15 weeks to the Veterans home via home-based clinical video teleconferencing (CVT).
  Interventions: Behavioral: CBCT-Home Based (CBCT-HB)
- CBCT-Office Based (CBCT-OB) (Active Comparator): Couples in CBCT-OB will receive 8 sessions of standardized Cognitive-Behavioral Conjoint Therapy (CBCT), a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning. The psychotherapy is administered over 8 to 15 weeks in-person in the therapist's office.
  Interventions: Behavioral: CBCT-Office Based (CBCT-OB)
- PTSD Family Education (PFE) (Active Comparator): Couples in the PFE condition will receive 8 sessions of standardized PTSD Family Education, a manualized psychoeducational program designed to help couples learn more about posttraumatic stress disorder and related difficulties. This psychotherapy is administered over 8 to 15 weeks and is delivered in-person in the therapist's office.
  Interventions: Behavioral: PTSD Family Education (PFE)

INTERVENTIONS:
Behavioral: CBCT-Home Based (CBCT-HB) — Couples in CBCT-HB will receive 8 sessions of standardized Cognitive-Behavioral Conjoint Therapy (CBCT), a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning. The psychotherapy is administered over 8 to 15 weeks to the Veterans home via home-based clinical video teleconferencing (CVT).
  Arms: CBCT-Home Based (CBCT-HB)
Behavioral: CBCT-Office Based (CBCT-OB) — Couples in CBCT-OB will receive 8 sessions of standardized Cognitive-Behavioral Conjoint Therapy (CBCT), a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning. The psychotherapy is administered over 8 to 15 weeks in-person in the therapist's office.
  Arms: CBCT-Office Based (CBCT-OB)
Behavioral: PTSD Family Education (PFE) — Couples in the PFE condition will receive 8 sessions of standardized PTSD Family Education, a manualized psychoeducational program designed to help couples learn more about posttraumatic stress disorder and related difficulties. This psychotherapy is administered over 8 to 15 weeks and is delivered in-person in the therapist's office.
  Arms: PTSD Family Education (PFE)

SUMMARY:
Untreated posttraumatic stress disorder (PTSD) is a costly condition associated with impairment in functioning across a host of psychosocial domains including occupational and academic functioning, marital and family functioning, parenting, and socialization. Impairment is not limited to Veterans with PTSD because the entire family is affected, particularly the Veteran's intimate partner. PTSD symptoms can produce negative effects on both members of the dyad. Despite the need for treatment, many Veterans and their families do not access PTSD-related services due to a number of barriers to accessing care (e.g., living in rural or remote areas where no specialty services exist, concerns about stigma around using mental health services, limited clinic hours to accommodate patient schedules). The objective of this study is to assess whether providing Cognitive-Behavioral Conjoint Therapy, in which PTSD symptoms and intimate relationship functioning are addressed, to Veterans and their romantic partners in their homes via clinical video teleconferencing leads to better outcomes compared to office based treatment.

DETAILED DESCRIPTION:
Anticipated Impact on Veterans' Healthcare: This project addresses the mental health and functioning needs of Veterans and their families by increasing the access to an established treatment using telemental health technology.

Project Background: Veterans and their families experience the deleterious effects of posttraumatic stress disorder (PTSD) and associated negative sequelae. PTSD is related to a variety of comorbid mental health symptomatology and psychosocial impairment, including high rates of intimate relationship problems which impact Veterans' recovery and functioning. Despite available couple-based interventions, barriers to care such as stigma regarding mental health treatment, travel time to receive care, and transportation costs, make it difficult for Veterans and their families to access specialty PTSD treatments necessary for rehabilitation. Home-based clinical video teleconferencing (CVT) delivers specialized mental health treatments to clients in the ease of their own home, which allows clinicians to directly observe the client's home environment and family milieu. Cognitive-Behavioral Conjoint Therapy (CBCT), a couple-based treatment designed to target PTSD symptoms and improve individual and relationship functioning, has shown evidence of improvements in clinical symptom outcomes in research conducted with Veterans and their partners.

Project Objectives: This is a 4-year randomized controlled trial. The primary objective of this study is to compare the clinical efficacy (PTSD symptoms, relationship distress, and functional impairment) of CBCT delivered via an office-based (CBCT-OB) or a home-based CVT (CBCT-HB) delivery modality to the PTSD Family Education control condition (PFE). In addition, this study will estimate and compare the difference in clinical efficacy between CBCT delivered via an office-based (CBCT-OB) or a home-based CVT (CBCT-HB) delivery modality if indicated by results of the primary objective. This study will also compare process outcomes (therapeutic alliance, enrollment and dropout rates, and treatment satisfaction) for CBCT-OB, CBCT-HB, and PFE.

Project Methods: Participants will be 180 intent-to-treat couples in which one partner is a PTSD-positive Veteran. Couples will be randomly assigned to receive treatment through one of the three treatment delivery modalities: CBCT-OB, CBCT-HB or PFE. Assessments will be conducted at baseline, mid- and post-treatment, and 3- and 6-months post-treatment. The primary outcome variables of clinical efficacy will be measures of PTSD symptom severity, relationship distress, and functional impairment. Secondary outcome variables include PTSD diagnostic status, self- reported PTSD symptoms, depression, anger, and relationship conflict. Additionally, primary process outcomes will include measures of treatment retention, attendance, therapeutic alliance, and treatment satisfaction. Variability in scores for each of the primary and secondary outcome measures will be examined individually in a series of separate multilevel models. The results will provide evidence that can be used to further increase the clinical efficacy, ease of access to, and utilization of specialty PTSD treatment to Veterans and their families.

ELIGIBILITY:
Inclusion Criteria:

* Be a Veteran (age 18 or older) with a current Diagnostic and Statistical Manual-5 (DSM-5) diagnosis of PTSD (as assessed by the CAPS) no less than 3 months after the index trauma occurred (to allow for potential natural recovery)
* Be on a stable psychoactive medication regimen for at least 2 months (if eligible)
* Be an intimate partner (age 18 or older) who is willing to participate in the intervention.
* Be randomized into any of the three treatment conditions
* Have assessment and treatment sessions audio recorded
* Agree not to receive other individual or conjoint psychotherapy for PTSD during the treatment portion of the study
* Consistent with home-based clinical trials and actual clinical practice
* Participants enrolled into the study will need to have access to internet via Digital Subscriber Line (DSL) or a cable provider in case they are randomized into the home-based condition.

  * The frequency of occurrence of no internet service will be tracked
  * If the PTSD-positive Veteran is currently receiving treatment at the VA, study staff will consult with their primary clinician prior to their inclusion in the study

Exclusion Criteria:

* Current substance dependence in either member of the couple not in remission for at least 3 months, as assessed by the Alcohol Use Disorders Identification Test (AUDIT)108 and Drug Abuse Screening Test (DAST)
* Any current uncontrolled psychotic disorder in either member of the couple
* Imminent suicidality or homicidality in either member of the couple
* Any severe cognitive impairment in either member of the couple
* Any perpetration of severe physical or sexual relationship aggression in the past year (as assessed by the Conflict Tactics Scale-2 [CTS-2]).

  * Participants who do not meet study criteria will be offered referrals to alternate services, as well as assistance in contacting the referral sites as needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A. Morland, PsyD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morland LA, Knopp KC, Khalifian CE, Macdonald A, Grubbs KM, Mackintosh MA, Becker-Cretu JJ, Sautter FJ, Buzzella BA, Wrape ER, Glassman LH, Webster K, Sohn MJ, Glynn SM, Acierno R, Monson CM. A randomized trial of brief couple therapy for PTSD and relationship satisfaction. J Consult Clin Psychol. 2022 May;90(5):392-404. doi: 10.1037/ccp0000731. PMID 35604746
- [Derived] Khalifian CE, Bosch J, Knopp K, Delay C, Sohn MJ, Morland LA. Adverse childhood experiences, mental health, and relationship satisfaction in military couples. J Fam Psychol. 2022 Jun;36(4):630-635. doi: 10.1037/fam0000952. Epub 2022 Jan 27. PMID 35084882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the recruitment period from October 2016 to March 2020, we received 706 referrals from the myriad of community-based outpatient clinics (CBOCs; e.g., VA Mission Valley Clinic), VA associated clinics (e.g., Family Mental Health), and self-referrals, typically from Veterans who see our study ads (both virtual and physical) in the La Jolla VA Main Hospital.
Groups:
- PTSD Family Education (PFE): Couples in the PFE condition will receive 8 sessions of standardized PTSD Family Education, a manualized psychoeducational program designed to help couples learn more about posttraumatic stress disorder and related difficulties. This psychotherapy is administered over 8 to 15 weeks and is delivered in-person in the therapist's office.
  PTSD Family Education (PFE): Couples in the PFE condition will receive 8 sessions of standardized PTSD Family Education, a manualized psychoeducational program designed to help couples learn more about posttraumatic stress disorder and related difficulties. This psychotherapy is administered over 8 to 15 weeks and is delivered in-person in the therapist?s office.
Period: Overall Study
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Started | 92 | 92 | 90
Y1 (Number of enrollment in Year 1 of study (March 2017-December 2017)) | 26 | 26 | 28
Y2 (Number of enrollment in Year 2 of study (2018)) | 34 | 32 | 34
Y3 (Number of enrollment in Year 3 of study (2019)) | 28 | 30 | 24
Y4 (Number of enrollment in Year 4 of study (January 2020-March 2020)) | 4 | 4 | 4
Veteran Total (Total number of veteran participants) | 46 | 46 | 45
Intimate Partner Total (Total number of intimate partners of veterans) | 46 | 46 | 45
Completed | 72 | 72 | 70
Not Completed | 20 | 20 | 20
Not completed — Separation of couple | 6 | 8 | 2
Not completed — Withdrawal by Subject | 6 | 6 | 4
Not completed — Scheduling issues | 2 | 4 | 7
Not completed — Childcare | 2 | 0 | 2
Not completed — Withdrawal by PI | 2 | 2 | 0
Not completed — Moved away | 2 | 0 | 0
Not completed — Not Primary Health Concern | 0 | 0 | 2
Not completed — Transportation issues | 0 | 0 | 1
Not completed — Other | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE) | Total
Number analyzed (Participants) | 92 | 92 | 90 | 274
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 85 | 87 | 76 | 248
  >=65 years | 7 | 5 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.37 (12.42) | 39.25 (12.45) | 43.89 (15.24) | 41.82 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 45 | 137
  Male | 46 | 46 | 45 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 33 | 29 | 93
  Not Hispanic or Latino | 60 | 58 | 58 | 176
  Unknown or Not Reported | 1 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 2 | 7
  Asian | 5 | 2 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 5 | 3 | 1 | 9
  Black or African American | 13 | 21 | 12 | 46
  White | 50 | 46 | 53 | 149
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 16 | 18 | 15 | 49
CAPS-5 [Mean (Standard Deviation); unit: units on a scale] — Clinician-Administered PTSD Scale (CAPS-5) for Diagnostic and Statistical Manual-5 (DSM-5) is a 30-item structured diagnostic interview that is considered the gold standard in PTSD assessment. It is designed to make a categorical PTSD diagnosis and provide measure of symptom severity. The structure corresponds to the DSM-5 criteria and can be administered by clinicians, clinical researchers, or appropriately trained paraprofessionals.
  *Score range: 0-80 with higher score indicating greater symptom severity Population: CAPS-5 was only administered to veteran IP participants (i.e., half the total sample), not their intimate partners.
  units on a scale
    number analyzed (Participants) | 46 | 46 | 45 | 137
    (all) | 38.5 (9.35) | 37.2 (9.95) | 36.9 (9.14) | 37.5 (9.44)
B-IPF [Mean (Standard Deviation); unit: units on a scale] — The Brief Inventory of Psychosocial Functioning (B-IPF) is a 7-item self-report questionnaire that assesses PTSD-related psychosocial functional impairment, an abridged version of the 80-item Inventory of Psychosocial Functioning questionnaire.
  *Score range: 0-100 with higher score indicating greater impairment Population: B-IPF was only administered to veteran IP participants (i.e., half the total sample), not their intimate partners.
  units on a scale
    number analyzed (Participants) | 46 | 46 | 45 | 137
    (all) | 42.0 (21.5) | 41.6 (21.8) | 39.8 (19.3) | 41.1 (20.8)
CSI [Mean (Standard Deviation); unit: units on a scale] — Couples Satisfaction Index (CSI) is a 32-item self-report questionnaire designed to measure one's satisfaction in a relationship.
  *Higher sum scores (range 0 to 161) represent higher relationship satisfaction. Population: Some missing data on this scale at baseline due to reasons such as participant failure to complete self-report measure, participant declined to answer, or assessor did not administer based on clinical judgment at the time of assessment.
  units on a scale
    number analyzed (Participants) | 89 | 92 | 83 | 264
    (all) | 102.9 (31.4) | 104.8 (35.9) | 111.9 (30.0) | 106.4 (32.7)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: The CAPS-5 is a 30-item clinician administered interview designed to diagnose current and lifetime PTSD and to assess PTSD symptom-severity over the past week. The interview assesses 20 DSM-5 PTSD symptoms as well as onset, duration, distress, and functional impact, overall validity, PTSD severity, and presence of dissociation. Prior to assessing symptoms, the clinical interviewer works with the patient to establish an index-trauma and each follow-up question focuses on symptoms as they relate to the index trauma.
  *Score range: 0-80 with higher score indicating greater symptom severity
Time Frame: Baseline
Population: Entire enrolled sample, Veteran partners only; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale | 38.456522 (1.3791780) | 37.239130 (1.4665958) | 36.933333 (1.3627068)

2. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: as for outcome 1
Time Frame: 1 Month Post Treatment
Population: Entire enrolled sample, Veteran partners only; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale | 25.400853 (2.0912490) | 25.949376 (2.0622709) | 31.697835 (2.0545996)
Statistical Analysis 1: Comparison: CBCT-Office Based (CBCT-OB) vs PTSD Family Education (PFE); Analyses were pooled across 50 imputed data sets. We used piecewise/spline mixed-effects regression models: one slope estimated from baseline to post (treatment impacts), with a separate slope estimated from post to 6-months (maintenance); Test type: Superiority; p = .016, Mixed-effects regression; Models included random intercepts; Slope = -3.216, Standard Error of Mean 1.300
Statistical Analysis 2: Comparison: CBCT-Home Based (CBCT-HB) vs PTSD Family Education (PFE); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .002, Mixed-effects regression; Models included random intercepts; Slope = -4.110, Standard Error of Mean 1.308
Statistical Analysis 3: Comparison: CBCT-Home Based (CBCT-HB) vs CBCT-Office Based (CBCT-OB); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .492, Mixed-effects regression; Models included random intercepts; Slope = -0.894, Standard Error of Mean 1.296

3. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: as for outcome 1
Time Frame: 3-Months Post Treatment
Population: Entire enrolled sample, Veteran partners only; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale | 24.483465 (2.2550249) | 24.647374 (2.2486121) | 30.361910 (2.2410544)

4. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: as for outcome 1
Time Frame: 6- Months Post Treatment
Population: Entire enrolled sample, Veteran partners only; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale | 25.225243 (2.3268567) | 24.869300 (2.3450681) | 28.281612 (2.2157577)

5. Primary Outcome: Couples Satisfaction Index (CSI)
Description: The Couples Satisfaction Index is a 32-item self-report survey assessing several domains of relationship satisfaction. Higher sum scores (range 0 to 161) represent higher relationship satisfaction.
Time Frame: Baseline
Population: Entire enrolled sample, both partners; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 92 | 92 | 90
score on a scale | 102.936782 (3.3421657) | 104.847826 (3.7405059) | 112.168689 (3.2376775)

6. Primary Outcome: Couples Satisfaction Index (CSI)
Description: as for outcome 5
Time Frame: Mid Treatment (Approximately week 5 of all treatment conditions)
Population: Entire enrolled sample, both partners; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 92 | 92 | 90
score on a scale | 103.004524 (3.8251803) | 108.112456 (4.1797505) | 114.748458 (3.5772543)

7. Primary Outcome: Couples Satisfaction Index (CSI)
Description: as for outcome 5
Time Frame: 1 Month Post Treatment
Population: Entire enrolled sample, both partners; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 92 | 92 | 90
score on a scale | 109.481289 (4.1068688) | 112.741213 (4.3721817) | 120.408861 (3.5479556)
Statistical Analysis 1: Comparison: CBCT-Office Based (CBCT-OB) vs PTSD Family Education (PFE); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .872, Mixed-effects regression; Models included random intercepts and included partners nested within couples; Slope = -0.352, Standard Error of Mean 2.172
Statistical Analysis 2: Comparison: CBCT-Home Based (CBCT-HB) vs PTSD Family Education (PFE); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .686, Mixed-effects regression; Models included random intercepts and included partners nested within couples; Slope = -0.931, Standard Error of Mean 2.296
Statistical Analysis 3: Comparison: CBCT-Home Based (CBCT-HB) vs CBCT-Office Based (CBCT-OB); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .798, Mixed-effects regression; Models included random intercepts and included partners nested within couples; Slope = -0.579, Standard Error of Mean 2.256

8. Primary Outcome: Couples Satisfaction Index (CSI)
Description: as for outcome 5
Time Frame: 3- Months Post Treatment
Population: Entire enrolled sample, both partners; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 92 | 92 | 90
score on a scale | 108.873270 (4.3020165) | 111.135788 (4.8525214) | 119.612750 (3.8630495)

9. Primary Outcome: Couples Satisfaction Index (CSI)
Description: as for outcome 5
Time Frame: 6- Months Post Treatment
Population: Entire enrolled sample, both partners; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 92 | 92 | 90
score on a scale | 109.384934 (4.1233647) | 110.919753 (4.7608962) | 118.410443 (3.9590245)

10. Primary Outcome: Inventory of Psychosocial Functioning (IPF)
Description: The Inventory of Psychosocial Functioning (IPF) is an 80-item self-report measure designed to assess multiple dimensions of functional impairment related to psychiatric disturbances. Higher sum scores (range 0 to 100) indicate more functional impairment.
Time Frame: Baseline
Population: Entire enrolled sample, Veteran partners only; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale | 50.1419 (3.53773) | 50.2336 (3.63994) | 47.5630 (3.42855)

11. Primary Outcome: Inventory of Psychosocial Functioning (IPF)
Description: as for outcome 10
Time Frame: Mid Treatment (Approximately week 5 of all treatment conditions)
Population: Entire enrolled sample, Veteran partners only; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale | 43.4390 (3.79594) | 43.0393 (3.68072) | 44.8664 (3.95252)

12. Primary Outcome: Inventory of Psychosocial Functioning (IPF)
Description: as for outcome 10
Time Frame: 1 Month Post Treatment
Population: Entire enrolled sample, Veteran partners only; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale | 33.2541 (4.09738) | 33.9657 (3.82502) | 34.0572 (3.88240)
Statistical Analysis 1: Comparison: CBCT-Office Based (CBCT-OB) vs PTSD Family Education (PFE); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .631, Mixed-effects regression; Models included random intercepts; Slope = -1.213, Standard Error of Mean 2.518
Statistical Analysis 2: Comparison: CBCT-Home Based (CBCT-HB) vs PTSD Family Education (PFE); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .560, Mixed-effects regression; Models included random intercepts; Slope = -1.461, Standard Error of Mean 2.495
Statistical Analysis 3: Comparison: CBCT-Home Based (CBCT-HB) vs CBCT-Office Based (CBCT-OB); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .922, Mixed-effects regression; Models included random intercepts; Slope = -0.248, Standard Error of Mean 2.536

13. Primary Outcome: Inventory of Psychosocial Functioning (IPF)
Description: as for outcome 10
Time Frame: 3- Months Post Treatment
Population: Entire enrolled sample, Veteran partners only; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale | 35.6696 (4.15061) | 33.6290 (4.37150) | 34.5942 (4.08413)

14. Primary Outcome: Inventory of Psychosocial Functioning (IPF)
Description: as for outcome 10
Time Frame: 6- Months Post Treatment
Population: Entire enrolled sample, Veteran partners only; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale | 38.3285 (4.15604) | 34.5207 (4.36232) | 37.2820 (4.10112)

15. Primary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: Client Satisfaction Questionnaire (CSQ) is an 8-item measure about satisfaction with treatment rated on a 4-point Likert scale. Higher mean scores (range 0 to 4) represent higher satisfaction with treatment services.
Time Frame: 1 Month Post Treatment
Population: Entire enrolled sample, both partners; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 92 | 92 | 90
score on a scale | 3.389157 (.1080726) | 3.423814 (.1029292) | 3.421993 (.1092805)

16. Primary Outcome: Working Alliance Inventory- Short Form (WAI-S)
Description: This adaptation of the Working Alliance Inventory- short form (WAI-S) includes 14 items assessing therapeutic alliance as reported by the patient on a 7-point Likert scale. Higher sum scores (14 to 98) represent higher patient-reported working alliance.
Time Frame: Approximately week 3 of all treatment conditions
Population: Entire enrolled sample, both partners; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 92 | 92 | 90
score on a scale | 67.039390 (1.3983512) | 71.116745 (1.3928316) | 68.748339 (1.6357681)

17. Primary Outcome: Working Alliance Inventory- Short Form (WAI-S)
Description: as for outcome 16
Time Frame: Approximately week 8 of all treatment conditions
Population: Entire enrolled sample, both partners; imputed using fully Bayesian model-consistent multiple imputation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 92 | 92 | 90
score on a scale | 72.099053 (1.3878994) | 73.882508 (1.4738266) | 75.647561 (1.4537812)

18. Secondary Outcome: PTSD Checklist-5 (PCL-5)
Description: The PCL-5 is a 20 item self report questionnaire assessing symptoms of PTSD based on DSM-V criteria. Scores range from 0 to 80, with higher scores representing more severe symptoms.
Time Frame: Baseline
Population: Entire enrolled sample, both partners, using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans | 50.3573 (2.39404) | 50.5211 (2.22140) | 51.2357 (2.20064)
  Intimate Partners | 16.5869 (2.09389) | 16.6637 (2.13649) | 15.6440 (1.94226)

19. Secondary Outcome: PTSD Checklist-5 (PCL-5)
Description: as for outcome 18
Time Frame: Mid Treatment (Approximately week 5 of all treatment conditions)
Population: Entire enrolled sample, both partners, using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans | 38.0555 (3.35830) | 40.1717 (3.38226) | 44.8501 (3.61442)
  Intimate Partners | 31.2492 (4.04086) | 25.7970 (3.86422) | 30.2030 (3.93086)

20. Secondary Outcome: PTSD Checklist-5 (PCL-5)
Description: as for outcome 18
Time Frame: 1 Month Post Treatment
Population: Entire enrolled sample, both partners, using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans | 34.1452 (3.75753) | 31.1537 (3.39480) | 42.1752 (3.53403)
  Intimate partners | 28.9042 (3.92662) | 25.2462 (3.54497) | 27.4718 (3.14068)

21. Secondary Outcome: PTSD Checklist-5 (PCL-5)
Description: as for outcome 18
Time Frame: 3- Months Post Treatment
Population: Entire enrolled sample, both partners, using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans | 36.2751 (3.66118) | 30.1964 (3.83395) | 38.3393 (3.43143)
  Intimate Partners | 27.5520 (4.20814) | 26.1153 (3.98684) | 28.9425 (4.09243)

22. Secondary Outcome: PTSD Checklist-5 (PCL-5)
Description: as for outcome 18
Time Frame: 6-Months Post Treatment
Population: Entire enrolled sample, both partners, using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans | 35.6725 (3.70946) | 31.0392 (3.71211) | 39.8824 (3.63766)
  Partners | 27.8900 (3.90941) | 25.1507 (3.94430) | 27.9336 (3.78858)

23. Secondary Outcome: Beck Depression Inventory-II (BDI-2)
Description: The BDI is a 21-item self report questionnaire assessing symptoms of depression. Scores range from 0 to 63, with higher scores representing more severe symptoms.
Time Frame: Baseline
Population: Entire enrolled sample, both partners, using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans | 29.2906 (2.01236) | 26.6096 (1.74223) | 26.7542 (1.91770)
  Intimate Partners | 11.3114 (1.32078) | 11.8069 (1.33799) | 11.4000 (1.48861)

24. Secondary Outcome: Beck Depression Inventory-II (BDI-2)
Description: as for outcome 23
Time Frame: Mid Treatment (Approximately Week 5 of all treatment conditions)
Population: Entire enrolled sample, both partners, using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans | 19.9002 (2.40992) | 20.4560 (2.22070) | 23.4512 (2.90633)
  Intimate Partners | 15.8047 (2.19033) | 12.4473 (2.63256) | 13.2118 (2.82790)

25. Secondary Outcome: Beck Depression Inventory-II (BDI-2)
Description: as for outcome 23
Time Frame: 1 Month Post Treatment
Population: Entire enrolled sample, both partners, using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans | 18.6926 (2.50075) | 15.6840 (2.42694) | 21.6229 (2.59271)
  Intimate Partners | 12.5802 (2.48624) | 11.6098 (2.09489) | 11.5033 (2.26777)

26. Secondary Outcome: Beck Depression Inventory-II (BDI-2)
Description: as for outcome 23
Time Frame: 3- Months Post Treatment
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans | 19.7016 (2.61738) | 15.6977 (2.59297) | 18.4080 (2.63802)
  Intimate Partners | 11.8226 (2.42731) | 11.4500 (2.28087) | 12.1826 (2.31299)

27. Secondary Outcome: Beck Depression Inventory-II (BDI-2)
Description: as for outcome 23
Time Frame: 6-Months Post Treatment
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans | 18.0075 (2.51420) | 14.9098 (2.42697) | 20.0467 (2.57977)
  Intimate Partners | 12.1675 (2.29771) | 11.5881 (2.08941) | 11.1593 (2.34132)

28. Secondary Outcome: State-Trait Anger Inventory (STAXI)
Description: The STAXI-2 is a self-report questionnaire assessing state and trait anger. The State subscale (15 items) ranges from 15 to 60, and the Trait subscale (10 items) ranges from 10 to 40, with higher scores representing more anger.
Time Frame: Baseline
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans - State subscale | 21.9205 (1.44069) | 23.3263 (1.66076) | 23.6691 (1.66970)
  Intimate Partners - State subscale | 16.5972 (.48672) | 16.5322 (.58332) | 16.3185 (.46291)
  Veterans - Trait subscale | 22.7246 (.85906) | 22.4783 (.76595) | 23.6012 (1.08541)
  Intimate Partners - Trait subscale | 15.9926 (.57623) | 17.3426 (.87470) | 16.2507 (.76938)

29. Secondary Outcome: State-Trait Anger Inventory (STAXI)
Description: as for outcome 28
Time Frame: Mid Treatment (Approximately week 5 of all treatment conditions)
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans - State subscale | 20.8798 (1.39310) | 20.5599 (1.49279) | 23.5422 (1.99174)
  Intimate Partners - State subscale | 19.0822 (1.19655) | 17.2434 (1.09043) | 17.7080 (1.27415)
  Veterans - Trait subscale | 19.5022 (1.03512) | 20.3355 (1.04492) | 21.6513 (1.32337)
  Intimate Partners - Trait subscale | 17.0778 (1.00838) | 17.0418 (.96957) | 16.8182 (1.02438)

30. Secondary Outcome: State-Trait Anger Inventory (STAXI)
Description: as for outcome 28
Time Frame: 1 Month Post Treatment
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans - State subscale | 19.6216 (1.51017) | 18.6260 (1.36216) | 22.0156 (1.57502)
  Intimate Partners - State subscale | 17.7897 (1.25246) | 17.8016 (1.21990) | 17.9761 (1.24466)
  Veterans - Trait subscale | 19.2848 (1.12873) | 19.0268 (1.11595) | 21.5299 (1.35408)
  Intimate Partners - Trait subscale | 16.4488 (1.13420) | 16.6423 (1.12928) | 16.4590 (1.01050)

31. Secondary Outcome: State-Trait Anger Inventory (STAXI)
Description: as for outcome 28
Time Frame: 3- Months Post Treatment
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans - Trait subscale | 18.7056 (1.20307) | 18.9492 (1.32233) | 20.5660 (1.37056)
  Intimate partners - Trait subscale | 15.9029 (1.22085) | 16.9785 (1.08067) | 16.7127 (1.14092)
  Veterans - State subscale | 20.5553 (1.69937) | 19.7572 (1.76798) | 20.0755 (1.48921)
  Intimate partners - State subscale | 17.8972 (1.23307) | 17.4860 (1.23456) | 18.8452 (1.25349)

32. Secondary Outcome: State-Trait Anger Inventory (STAXI)
Description: as for outcome 28
Time Frame: 6-Months Post Treatment
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans - State subscale | 19.9870 (1.37717) | 20.0932 (1.67819) | 20.8182 (1.31146)
  Intimate Partners - State subscale | 17.5131 (1.26957) | 17.2149 (1.19453) | 17.7645 (1.18880)
  Veterans - Trait subscale | 18.4906 (1.07693) | 18.9074 (1.25158) | 19.7710 (1.14792)
  Intimate Partners - Trait subscale | 16.0526 (1.22372) | 16.2891 (1.09040) | 16.0928 (1.09770)

33. Secondary Outcome: Conflict Tactics Scale Short Form- (CTS-2S)
Description: 20-item self-report inventory yielding 5 scales. Most widely used measure of its kind. Scores on the Psychological Aggression and Negotiation subscales range from 0 to 24, with higher scores representing more Psychological Aggression and more Negotiation.
Time Frame: Baseline
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans - Psychological aggression subscale | 8.1739 (.58591) | 8.5217 (.63149) | 7.8444 (.55592)
  Intimate Partners - Psychological aggression subscale | 8.9130 (.50296) | 7.8696 (.60242) | 7.5778 (.68423)
  Veterans - Negotiation subscale | 17.5000 (.74129) | 18.2174 (.76828) | 18.7111 (.65568)
  Intimate Partners - Negotiation subscale | 18.4348 (.61042) | 17.7609 (.70689) | 17.4889 (.86551)

34. Secondary Outcome: Conflict Tactics Scale Short Form- (CTS-2S)
Description: as for outcome 33
Time Frame: Mid Treatment (Approximately week 5 of all treatment conditions)
Population: Enrolled sample only, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans - Psychological aggression subscale | 4.3120 (.72809) | 4.8690 (.64106) | 3.6182 (.70126)
  Intimate Partners - Psychological aggression subscale | 4.2366 (.72491) | 4.6851 (.65959) | 3.5465 (.65402)
  Veterans - Negotiation subscale | 13.6238 (1.02718) | 13.7363 (.89228) | 14.6018 (.91310)
  Intimate Partners - Negotiation subscale | 13.9197 (1.01009) | 12.9316 (.95512) | 14.2217 (.89814)

35. Secondary Outcome: Conflict Tactics Scale Short Form- (CTS-2S)
Description: as for outcome 33
Time Frame: 1 Month Post Treatment
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans - Psychological aggression subscale | 4.1295 (.71564) | 4.0524 (.68690) | 3.4079 (.63721)
  Intimate Partners - Psychological aggression subscale | 3.5965 (.65219) | 4.7797 (.65758) | 3.7661 (.68853)
  Veterans - Negotiation subscale | 14.9523 (.99330) | 14.6470 (.99507) | 14.9224 (.94777)
  Intimate Partners - Negotiation subscale | 15.3302 (.90193) | 14.9261 (1.03747) | 14.3585 (1.11890)

36. Secondary Outcome: Conflict Tactics Scale Short Form- (CTS-2S)
Description: as for outcome 33
Time Frame: 3- Months Post Treatment
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans - Psychological aggression subscale | 4.0795 (.69410) | 4.0335 (.69447) | 3.7106 (.60643)
  Intimate partners - Psychological aggression subscale | 3.7899 (.71769) | 4.5018 (.69773) | 3.8952 (.66721)
  Veterans - Negotiation subscale | 14.7853 (1.00807) | 14.8986 (1.07100) | 14.3893 (1.11230)
  Intimate Partners - Negotiation subscale | 15.0919 (1.03404) | 14.6806 (1.04556) | 14.3492 (1.02322)

37. Secondary Outcome: Conflict Tactics Scale Short Form- (CTS-2S)
Description: as for outcome 33
Time Frame: 6-Months Post Treatment
Population: Entire enrolled sample, both partners; using multiply imputed data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
Number analyzed (Participants) | 46 | 46 | 45
score on a scale
  Veterans - Psychological aggression subscale | 4.2911 (.79419) | 4.1617 (.72540) | 3.1872 (.65897)
  Intimate Partners - Psychological aggression subscale | 3.9574 (.68440) | 4.5597 (.71441) | 3.5832 (.67381)
  Veterans - Negotiation subscale | 14.4958 (1.06696) | 13.9513 (1.15916) | 13.4718 (1.06347)
  Intimate Partners - Negotiation subscale | 15.7043 (.97081) | 13.6076 (1.13738) | 15.0468 (1.10333)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected for up to 1 year since the date of baseline.
Description: Clinicaltrials.gov definition is consistent with definition used for the duration of the study.
Arm/Group | CBCT-Home Based (CBCT-HB) | CBCT-Office Based (CBCT-OB) | PTSD Family Education (PFE)
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/92 | 0/92
Other Adverse Events (participants affected / at risk) | 8/92 | 14/92 | 14/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBCT-Home Based (CBCT-HB) (N=92) | CBCT-Office Based (CBCT-OB) (N=92) | PTSD Family Education (PFE) (N=90)
Emergency room visit (General disorders) | 2 (2) | 1 (1) | 3 (3) — Unrelated to study. Same-day discharge from ER.
Hospitalization (General disorders) | 3 (3) | 3 (3) | 2 (2) — Unrelated to study
Surgery (General disorders) | 1 (1) | 1 (1) | 0 (0) — Unrelated to study
APC Report (Social circumstances) | 1 (1) | 1 (1) | 3 (3) — Unrelated to study. Mandated report.
CPS Report (Social circumstances) | 0 (0) | 2 (2) | 0 (0) — Unrelated to study. Mandated report.
Police visit (Investigations) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study. One incident where police visited participant's home due to noise complaint from domestic argument.
Protocol Deviation (Investigations) | 1 (1) | 1 (1) | 0 (0) — Total of 2 protocol deviations reported (unrelated to study). 1. Participant incarcerated during therapy due to parole violation. 2. Participant escorted by VA police for psychiatric evaluation for damaging the wall.
Protocol Deviation-COVID-19 (General disorders) | 0 (0) | 4 (10) | 6 (12) — Unrelated to study. Due to the COVID-19 pandemic shutdown in San Diego, a total of 10 participants (5 couples) received home-based telehealth treatment despite being randomized to an office-based condition.

LIMITATIONS AND CAVEATS:
Study exclusion criteria (e.g., recent aggression, suicidality) may have excluded couples with more severe pathology. All measures except for the CAPS-5 were self-reported measures, introducing potential bias in reporting. This study involved significant administrative support for telehealth procedures; not all VA clinical settings will include these administrative supports, which may reduce generalizability of our results to standard clinical care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT02720016/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT02720016/SAP_001.pdf